CLINICAL TRIAL: NCT00108992
Title: Efficacy and Safety of Topical Diclofenac Combined With Oral Diclofenac in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nuvo Research Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEN-03-112
Record Dates: First submitted 2005-04-21; First posted 2005-04-22 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Osteoarthritis, Knee
Keywords: topical NSAID; topical diclofenac
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Diclofenac

INTERVENTIONS:
Drug: Diclofenac, topical

SUMMARY:
Oral non-steroidal anti-inflammatory drugs (NSAIDs) are a recommended treatment for the symptoms of osteoarthritis of the knee. However, NSAIDs may cause a range of negative side effects, including stomach pain, heartburn, bleeding stomach ulcer, and liver or kidney abnormality. A topical NSAID may relieve pain and other symptoms of osteoarthritis of the knee, while minimizing the side effects common to oral NSAIDs. The purpose of this study is to determine the safety and effectiveness of a topical NSAID when used alone or when combined with an oral NSAID in the treatment of osteoarthritis of the knee.

DETAILED DESCRIPTION:
During this 12-week study, patients will visit the study clinic 5 times. At the screening visit, the patient's demographic information, medical and medication history will be recorded and a physical examination performed. After washout of all NSAIDs/other analgesic medication, the patient will return for the baseline visit. During the treatment phase of the study, the patient will apply a topical solution to his/her osteoarthritic knee and take an oral study tablet. The patient may randomly receive active treatment with topical diclofenac, oral diclofenac, both, or neither (placebo). Follow-up clinic visits are conducted at 4, 8 and 12 weeks. Routine laboratory analyses are done at baseline, 4 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the knee, verified radiographically
* Moderate flare of pain in the knee after washout of stable therapy
* If female, non-pregnant
* Ability to swallow moderately-sized tablets

Exclusion Criteria:

* Secondary osteoarthritis of the knee
* Major knee surgery at any time, or minor knee surgery in previous year
* Severe uncontrolled heart, liver or kidney disease
* Ulcer or bleeding from the stomach
* Corticosteroid use
* Fibromyalgia
* Skin disorder of the knee

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 2004-02; Study Completion 2005-09

PRIMARY OUTCOMES:
pain
physical function
patient overall health assessment

SECONDARY OUTCOMES:
stiffness
patient global assessment

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Coastal Clinical Research, Mobile, Alabama
  - Redpoint Research, Phoenix, Arizona
  - OMC Clinical, Beverly Hills, California
  - Associated Pharmaceutical Research, Buena Park, California
  - Med Investigators, Fair Oaks, California
  - Desert Medical Advances, Palm Desert, California
  - Boling Clinical Trials, Upland, California
  - Tampa Bay Medical Research Inc., Clearwater, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Medisphere Medical Research, Evansville, Indiana
  - Synergy Medical Education Alliance, Saginaw, Michigan
  - Redrock Research Center, Las Vegas, Nevada
  - Partners in Primary Care, Voorhees Township, New Jersey
  - Camp Hill Clinical Research Center, Camp Hill, Pennsylvania
  - Primary Physicians Research, Pittsburgh, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Research Associates, Nashville, Tennessee
  - Research Across America, Dallas, Texas
  - Sam Clinical Research Center, San Antonio, Texas
  - Hamptom Roads Center for Clinical Research, Norfolk, Virginia
  - National Clinical Research, Richmond, Virginia